CLINICAL TRIAL: NCT02861378
Title: Reversing the Effects of 2% Lidocaine: A Randomized Controlled Trial
Brief Title: Reversing the Effects of 2% Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-3515
Record Dates: First submitted 2016-06-22; First posted 2016-08-10 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Soft Tissue Anaesthesia
Keywords: anaesthesia, dental; lidocaine
MeSH Terms: interventions — Phentolamine; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phentolamine mesylate (Experimental): Once anesthesia is confirmed, subjects in the Phentolamine mesylate group will receive 1 injection of 1ml of a solution containing 0.24 mg of phentolamine mesylate in the same site that was previously anaesthetized (not as a part of the study).
  Interventions: Drug: Phentolamine mesylate
- Water (Placebo Comparator): Once anaesthesia is confined, the subjects in the water group will receive 1 injection of 1 ml of sterile physiological water in the same site that was previously anaesthetized (not as a part of the study).
  Interventions: Drug: Water

INTERVENTIONS:
Drug: Phentolamine mesylate — Injection of 1ml at lidocaine injection site
  Other Names: OraVerse
  Arms: Phentolamine mesylate
Drug: Water — Injection of 1ml of physiologic saline water at injection site
  Arms: Water

SUMMARY:
Dental procedures often require the use of local anesthesia. The effects of the anesthesia usually linger for some time after the dental procedure is completed which can lead to discomfort and occasionally injury from lip/tongue biting. Clinical trials have shown phentolamine mesylate (OraVerse) to be effective at reducing the amount of time to reversal of local anesthesia compared to sham injections. However, no trials have been conducted comparing phentolamine mesylate to a true control injection. Such trials are needed in order to definitively show that it is the phentolamine mesylate itself that is causing the reduction in anesthesia rather than a dilution effect.

The objective of the proposed research is to conduct a pilot-scale randomized clinical trial evaluating the difference in time required to the return of normal soft-tissue sensation and function in participants who had received an inferior alveolar nerve block (using 2% Lidocaine 1:100,000 epinephrine), followed by an injection with either 1) OraVerse (phentolamine mesylate) or 2) sterile physiological water (control).

The study population will comprise dentistry and dental hygiene students of the second year classes at Dalhousie University, Halifax, NS, Canada. This study population has been chosen because these students usually practice dental anesthesia on each other as a part of a course on local anesthesia.

This proposed pilot scale study will be a double-blind controlled trial using parallel groups. As part of their usual anaesthesia course, the dental and dental hygiene students will be practicing their inferior alveolar nerve injections on one another using 2% Lidocaine 1:100,000 epinephrine. Students who decide to participate in the study will be randomly assigned to one of two groups: Group 1 will receive an injection of OraVerse (treatment group), while Group 2 will receive an injection of sterile physiological water (control group). The time required to the return of soft-tissue sensation and function will be assessed using a questionnaire.

DETAILED DESCRIPTION:
The research will be conducted at the Dalhousie University Dental Clinic. As part of their anaesthesia clinical course, students enrolled in the second year of the dentistry and dental hygiene programs practice different anesthesia techniques on each other during a planned hands-on training activity. The research study will take place during the same day. Participants who meet the eligibility criteria and consent to participate will be randomly assigned to one of two groups. Following anesthesia obtained as a part of their hands-on training session, subjects allocated to Group 1 will receive 1ml of phentolamine mesylate following anesthesia, while subjects allocated to Group 2 will receive 1ml of sterile physiological water.

Phase 1, Both Groups:

1. Subjects will be trained to use the Assessment of Anesthesia questionnaire
2. Following training, subjects will perform baseline assessments of their lip and tongue numbness (should be normal).
3. Prior to anaesthesia is given, vital signs will be recorded. Blood pressure, respiratory rate and pulse will all be recorded.
4. Topical anesthetic, 20% benzocaine, will be applied to the injection site for 3 minutes. Subjects will be given a standard inferior alveolar nerve block injection, with aspiration before injection, using 1ml of 2% lidocaine with 1:100,000 epinephrine from the student they are teamed with. This step is not part of the study; it is done as part of their clinical anesthesia course.
5. Soft tissue anaesthesia will be self-assessed, by using finger tapping and palpation, to ensure profound anesthesia. The second phase (OraVerse or water) will not take place before profound anesthesia has been achieved. The anesthetic outcome will be considered a failure if the participant does not report anesthesia of the lower lip within 10 minutes.
6. If profound anesthesia is achieved within 10 minutes, subjects will proceed to phase 2. If profound anesthesia is not achieved within 10 minutes subjects will be withdrawn from the study. Subjects who are withdrawn from the study will continue with their standard training protocol which is to receive a re-injection of anesthetic. A withdrawal form will be used by Dr. Flood to record the occurrence of anesthesia failures. This form will also record reasons for withdrawals, should any occur for different reasons.

Phase 2 Group 1: Phentolamine Mesylate After anesthesia is confirmed, subjects in Group 1 will receive an injection of 1ml of a solution containing 0.24mg of phentolamine mesylate in the same site previously injected with anaesthetic solution. Dr. Brittany Flood will give the injection to ensure consistency.

Group 2: Water After anesthesia is confirmed, subjects in Group 2 will receive an injection of 1ml of sterile physiological water in the same site previously injected with anesthetic solution. Dr. Brittany Flood will give the injection to ensure consistency.

Phase 3 Vital signs will be taken immediately after injection, by their student partner, and all students will be monitored for 30 minutes. During the monitoring period, the participants will self-assess their anesthesia, using the Assessment Of Anesthesia questionnaire. This self-assessment will be done every ten minutes until soft-tissues revert to their normal state. After the 30 minute monitoring period participants will be free to leave the clinic, taking the questionnaire with them but will continue to check for anesthesia every 10 minutes until tissue sensation and function return to normal. Students will be instructed to return the forms to the office of the Research Development Officer.

The Case Report Forms will include the following:

* Assessment Of Anesthesia questionnaire: self-assessment of state of soft-tissue anesthesia
* Subject Eligibility Checklist: inclusion/exclusion criteria
* Consent form
* Participant Identification allocation Log (centrally kept): Participant study ID and chart number
* Treatment Group Allocation Log (centrally kept): Participant study ID and treatment group ('A' or 'B')
* Withdrawal information
* Adverse Event form

Recruitment and reversal injections will be done by Dr. Brittany Flood, who is a licensed dentist currently enrolled as a student in the Masters of Periodontics program at Dalhousie University Faculty of Dentistry. Dr. Pierre-Luc Michaud who is a dentist and full-time assistant professor at Dalhousie Dentistry will supervise the project and perform data analysis. He will not be involved in recruitment and will not be present during the clinical phase of the study. Dr. Brittany Flood is not in a position of authority with the dental or dental hygiene students and will therefore be the only research member working directly with the participants. She will be the only research team member aware of who has volunteered to be in the study.

Two weeks before the anesthesia session, the potential participants will be given a thirty minute presentation, followed by a question and answer session. On the evening of the anesthesia course session, the initial numbness assessment (2 minutes) and reversal injection (5 minutes) will be the only clinical time required from participants in the study, as the other manipulations (vital signs monitoring and 30 minutes post-injection waiting-time period before leaving) are a standard part of their course. Following the clinical portion, participants will be free to leave the clinic but will continue to check for anesthesia every 10 minutes and then fill out a short questionnaire when sensation and function return to normal (to record duration of soft-tissue anesthesia). The duration of anesthesia could take between 1 and 2.5 hours, depending in which group the participant is.

This study is a randomized double-blind study. The Research Development Officer of the Faculty of Dentistry will be responsible for the randomization procedure. A computerized random number generator will be used to generate six randomly permuted blocks, with a block size of six. Within each block, an equal number of subjects will be allocated to the two treatment groups ('A' or 'B'). These will refer to either OraVerse group or Control group, but the Research Development Officer will withhold the information until the statistical analyses are completed. She will however give a copy to the supervisor of the anesthesia training session (who is not involved in the study) so that the information on what was injected could be quickly accessed during the hands-on if required and to appropriately fill participants' clinical chart. The allocations will be placed in sequentially numbered (01 through 36), opaque, sealed envelopes (referring to participants' ID) to be opened at the time of participant's reversal injection. The treatment group (A or B) randomly assigned for each participant will be recorded in the Treatment Group Allocation Log. The syringes will be marked as 'A' or 'B'; the person injecting (Dr. Brittany Flood) will not know which contains OraVerse (PM) and which contains water. As previously discussed, the anesthetic course supervisor will however have the information as a safety measure and to appropriate fill the patients' chart. To ensure continuous blinding of allocation, the randomization code will be kept secret by the Research Development Officer until after data analysis. Only the participant study ID will be used to label the subject's case report forms. Only the Participant Identification allocation Log could associate the participant ID with the patients' chart number, but this file will be kept centrally during the study time.

ELIGIBILITY:
Inclusion Criteria:

Students of the Dalhousie University Dental Clinic who are:

* Age 18 and over
* Capable of providing informed consent

Exclusion Criteria:

* Subjects with a medical history that contraindicates the use of epinephrine.
* Subjects who have taken an opioid or an opioid-like analgesic within 24 hours of the anesthesia session.
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time to return of normal soft tissue sensation and function | Every 10 minutes, from the injection of reversing agent or placebo until return to normal soft tissue sensation and function (up to 4 hours)
  Soft tissue anesthesia will be assessed using the Assessment of Anesthesia questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Luc Michaud, MSc, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University Faculty of Dentistry, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only in a publication in a dental journal

REFERENCES:
- [Derived] Michaud PL, Flood B, Brillant MS. Reversing the effects of 2% Lidocaine: A randomized controlled clinical trial. J Dent. 2018 May;72:76-79. doi: 10.1016/j.jdent.2018.03.009. Epub 2018 Mar 20. PMID 29571953
- See also: Dalhousie University Faculty of Dentistry Web Site — http://www.dal.ca/faculty/dentistry.html